CLINICAL TRIAL: NCT07264101
Title: Validity And Reliability Of The Four Square Step Test In Individuals With Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeynal Yasacı, Doctor lecturer, Inonu University
Other Study IDs: 1001
Record Dates: First submitted 2025-11-20; First posted 2025-12-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis (RA); Four Square Step Test (FSST); Balance
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis Group: Participants will consist of adult individuals aged 18-65 years with a diagnosis of rheumatoid arthritis based on the ACR/EULAR classification criteria. Clinical assessments will include the Four Square Step Test (FSST), Berg Balance Scale, Mini-BESTest, handgrip strength using a dynamometer. Disease activity (DAS28), pain intensity, quality of life, and history of falls will also be recorded. This study is purely observational and cross-sectional in nature, and no therapeutic intervention will be applied to participants.

SUMMARY:
This cross-sectional observational study aims to evaluate the validity and reliability of the Four Square Step Test (FSST) in individuals with rheumatoid arthritis. In addition, the study will investigate the associations between FSST performance and clinical parameters including disease activity, quality of life, pain, and muscle strength.

All assessments will be conducted according to a pre-defined standardized protocol. The order of measurement tools will be randomized to minimize potential bias, and sufficient rest intervals will be provided between tests to prevent fatigue and performance effects.

Participants will include individuals aged 18-65 years with a diagnosis of rheumatoid arthritis according to the ACR/EULAR 2010 classification criteria, who have been followed for at least 6 months, have had no major changes in treatment regimen in the last 4 weeks (e.g., initiation or change of DMARDs/biologics, high-dose steroid increase), can walk at least 10 meters independently, have a Mini-Mental State Examination score of 24 or higher, and are able to follow verbal instructions in Turkish to comply with study procedures.

Appropriate statistical methods will be applied to assess validity, reliability, and associations between FSST and clinical parameters.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, autoimmune connective tissue disease that affects approximately 0.5-1% of the global population. The disease is characterized by symmetrical joint pain, swelling, and restricted mobility. Synovial inflammation in its pathogenesis leads to structural damage, cartilage erosion, joint deformities, and irreversible functional impairments. Beyond joint involvement, RA significantly affects daily living activities, work capacity, and overall quality of life through its impact on the musculoskeletal system. Muscle weakness, reduced joint range of motion, and impaired proprioception occurring during the disease process particularly compromise lower extremity function and contribute to impaired postural control. Consequently, balance deficits, an increased risk of falls, and fall-related injuries are observed more frequently in individuals with RA compared to the healthy population.

Balance is generally divided into static and dynamic balance. Static balance refers to the ability to maintain the center of mass within the base of support while standing still, whereas dynamic balance denotes the ability to sustain the center of mass safely and in a controlled manner within the base of support during movement. In RA, balance impairments become especially evident in daily activities such as walking, changing direction, and climbing stairs. These difficulties elevate fall risk and adversely influence both physical independence and social participation.

Several assessment tools have been developed to evaluate balance in RA. The Berg Balance Scale (BBS), Tinetti Balance Test, Timed Up and Go Test (TUG), and Mini-BESTest are among the most widely used instruments in this field. However, many of these tools require lengthy administration, specialized equipment, or advanced clinical expertise. Such limitations can complicate rapid patient assessment, particularly in busy outpatient clinical settings.

The Four Square Step Test (FSST) is a practical assessment that can be administered within a short period of time using simple materials, measuring an individual's ability to step in multiple directions. The reliability and validity of FSST have been established in various clinical populations, including those with ankle injuries, hemophilia, cerebral palsy, Duchenne muscular dystrophy, Down syndrome, hip arthroplasty, and anterior cruciate ligament reconstruction. Nevertheless, no validity and reliability study of the FSST has yet been conducted in individuals with RA.

The primary objective of this study is to determine the validity and reliability of the Four Square Step Test (FSST) in individuals with rheumatoid arthritis. The secondary objective is to examine the relationship between FSST outcomes and clinical indicators such as disease activity, quality of life, pain and muscle strength.

First, demographic and clinical data of all participants will be collected, including age, height, weight, smoking and alcohol consumption, dominant side, use of assistive devices, age at diagnosis, comorbidities, medications, and history of falls within the past 1-2 years. Body mass index (BMI) will be calculated.

All analyses will be conducted as two-tailed, with a significance level set at α = 0.05, and results will be reported with 95% confidence intervals. The distribution of continuous variables will be assessed using the Shapiro-Wilk test. Normally distributed variables will be presented as mean ± standard deviation, while non-normally distributed variables will be reported as median values. Categorical variables will be presented as frequency (percentage).

The relationships between FSST time and the scores of the Berg Balance Scale (BBS) and Mini-BESTest will be examined using Pearson's or Spearman's correlation coefficients, depending on data distribution. The predictive ability of FSST for poor balance status will be evaluated with receiver operating characteristic (ROC) curve analysis, and results will be reported in terms of area under the curve (AUC), sensitivity, specificity, Youden's index, and optimal cutoff values.

Test-retest reliability will be determined using the intraclass correlation coefficient (ICC[3,1]) based on repeated FSST measurements performed by the same rater. Measurement error and minimal detectable change will be calculated as follows: SEM = SD × √(1 - ICC) and MDC95 = SEM × 1.96 × √2. Agreement between repeated measures will be illustrated using Bland-Altman plots (mean bias and ±1.96 SD limits).

Comparisons of FSST times between clinical subgroups (e.g., disease activity level, history of falls) will be performed using independent-samples t-test/ANOVA if normality assumptions are met, or Mann-Whitney U/Kruskal-Wallis tests otherwise. Effect sizes will be reported as Hedges' g, r, and η²/partial η².

Reporting will follow the STROBE guidelines for observational cross-sectional studies.

The sample size was calculated using the G*Power software with α = 0.05 and 1-β = 0.80. Previous studies have reported that the FSST demonstrates moderate to high levels of validity in different clinical populations. For example, in patients with hip osteoarthritis and total hip arthroplasty, correlations between FSST and other balance scales were found to range between r = 0.60 and r = 0.70. In individuals with total knee arthroplasty, FSST was reported to correlate with the TUG at r = 0.65 and with the HSS at r = -0.40. Furthermore, studies conducted in populations with hemophilia and Parkinson's disease indicated excellent reliability of FSST and modified FSST, with ICC values approximately between 0.96 and 0.99. Such studies have typically been conducted with sample sizes ranging from 17 to 28 participants.

In light of these findings, it was determined that including approximately 40 participants in the present study would be sufficient to ensure adequate statistical power for the planned validity analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Diagnosis of rheumatoid arthritis according to ACR/EULAR 2010 criteria
* No major changes in treatment regimen (e.g., initiation or modification of DMARDs/biologics, high-dose steroid increase) within the last 4 weeks
* Ability to walk at least 10 meters without assistance
* Mini-Mental State Examination (MMSE) score ≥ 24
* Ability to understand and follow instructions in Turkish

Exclusion Criteria:

* Participants who cannot understand or follow verbal instructions in Turkish
* Participants with a history of neurological, vestibular, or serious orthopedic disease
* Participants whose physical participation is limited due to acute infection or systemic disease
* Participants who have had lower extremity surgery or a history of serious injury within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 18-65 years with rheumatoid arthritis (RA) will be included in this study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Four Square Step Test (FSST) | Two assesstment ( one at baseline and one in the afternoon)
  The Four Square Step Test (FSST) is used to assess dynamic balance, specifically the ability to rapidly step over obstacles and change direction in a clinical setting. FSST is a quick and easily administered test that evaluates an individual's capacity to step in multiple directions over low obstacles. Four squares are created by intersecting lines at right angles, with each side approximately 90 cm in length. Low obstacles of 2.5 cm height are placed along the square boundaries. The participant starts in the lower-left square with feet together. In the first phase, the participant steps clockwise through each square-forward, right, backward, and left-returning to the starting position. The same sequence is then repeated counterclockwise. Participants must step into each square with both feet. After one practice trial, the test is performed twice, and completion times are recorded in seconds. The fastest time is considered the FSST score, with lower times indicating better dynamic bal

SECONDARY OUTCOMES:
Disease Activity Score-28 (DAS-28) | Baseline (First assessment)
  DAS28 is a widely used instrument for evaluating disease activity in individuals with rheumatoid arthritis. This index incorporates the number of tender and swollen joints out of 28, the patient's self-assessment of general health using a 100-mm visual analog scale (VAS), and acute-phase reactants, including erythrocyte sedimentation rate (ESR, mm/h) or C-reactive protein (CRP, mg/L). The resulting total score provides a quantitative measure of disease activity, with lower scores indicating remission and higher scores reflecting active disease
Numeric Rating Scale (NRS) | Baseline (First assesstment)
  The NRS is a unidimensional measure of pain intensity commonly used in adults. Multiple versions exist, but the 11-point scale (0-10) is the most widely employed. Patients are asked to select a number that best represents their pain intensity, where 0 indicates no pain and 10 represents the worst imaginable pain experienced over the past 24 hours.
Rheumatoid Arthritis Quality of Life (RAQoL) scale | Baseline (First assesstment)
  The Rheumatoid Arthritis Quality of Life (RAQoL) questionnaire is a disease-specific self-report instrument designed to assess quality of life in individuals with rheumatoid arthritis. The scale consists of 30 items with "yes/no" response options. Each "yes" response is scored as 1 point and each "no" response as 0 points, resulting in a total score ranging from 0 to 30. Lower scores indicate better quality of life, whereas higher scores reflect greater impairment in quality of life.
Mini-Balance Evaluation Systems Test (Mini-BESTest) | Baseline (First assesstment)
  The Mini-Balance Evaluation Systems Test (Mini-BESTest) is designed to assess dynamic balance using 14 items organized into four subscales: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. Each item is scored on a 3-point ordinal scale, with 0 indicating inability or need for assistance and 2 representing normal function. Total scores range from 0 to 28. Two items are evaluated for both the right and left sides, and only the lower score is included in the total score calculation.
Berg Balance Test(BBS) | Baseline ( First assessment)
  The Berg Balance Scale (BBS) is a balance assessment tool that evaluates an individual's ability to maintain stability while performing 14 functional tasks commonly encountered in daily activities. Each item is rated on a 5-point ordinal scale ranging from 0 to 4, where 0 indicates inability to perform the task and 4 represents the ability to complete the task independently. The maximum possible total score is 56. Administration of the test typically requires approximately 15-20 minutes.
Baseline Hydraulic Hand Dynamometer | Baseline (First assesstment)
  Participants are seated upright on a chair with their feet supported. The tested upper extremity is positioned with the shoulder in adduction and neutral rotation, the elbow at 90° flexion, the forearm in neutral position, and the wrist at 0-30° extension and 0-15° ulnar deviation. Participants are instructed to place their fingers around the dynamometer handle and squeeze with maximal force. The test is repeated three times, and the highest value obtained is used for analysis.
5 Times Sit To Stand Test (5TSTS) | Baseline (First assesstment)
  To assess quadriceps muscle strength and functional lower limb strength, the Five Times Sit-to-Stand Test (5TSTS) will be used.
  In the 5TSTS, participants are instructed to stand up and sit down five times as quickly as possible. A stopwatch is started with the command "start" and stopped upon completion of the fifth full standing position.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynal Yasacı, Principal Investigator — Inonü University
Locations (1):
- Inonu University Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant data will be securely stored by the investigators and may be shared with authorized personnel if deemed necessary, in accordance with applicable privacy regulations.

REFERENCES:
- [Background] Vilarinho R, Montes AM, Noites A, Silva F, Melo C. Reference values for the 1-minute sit-to-stand and 5 times sit-to-stand tests to assess functional capacity: a cross-sectional study. Physiotherapy. 2024 Sep;124:85-92. doi: 10.1016/j.physio.2024.01.004. Epub 2024 Jan 20. PMID 38875841
- [Background] Du W, Cornett KMD, Donlevy GA, Burns J, McKay MJ. Variability between Different Hand-Held Dynamometers for Measuring Muscle Strength. Sensors (Basel). 2024 Mar 14;24(6):1861. doi: 10.3390/s24061861. PMID 38544123
- [Background] Zonzini Gaino J, Barros Bertolo M, Silva Nunes C, de Morais Barbosa C, Sachetto Z, Davitt M, de Paiva Magalhaes E. Disease-related outcomes influence prevalence of falls in people with rheumatoid arthritis. Ann Phys Rehabil Med. 2019 Mar;62(2):84-91. doi: 10.1016/j.rehab.2018.09.003. Epub 2018 Sep 29. PMID 30278237
- [Background] Wagner S, Bring A, Asenlof P. Construct validity of the Mini-BESTest in individuals with chronic pain in specialized pain care. BMC Musculoskelet Disord. 2023 May 17;24(1):391. doi: 10.1186/s12891-023-06504-9. PMID 37198616
- [Background] Tijhuis GJ, de Jong Z, Zwinderman AH, Zuijderduin WM, Jansen LM, Hazes JM, Vliet Vlieland TP. The validity of the Rheumatoid Arthritis Quality of Life (RAQoL) questionnaire. Rheumatology (Oxford). 2001 Oct;40(10):1112-9. doi: 10.1093/rheumatology/40.10.1112. PMID 11600740
- [Background] Robinson CL, Phung A, Dominguez M, Remotti E, Ricciardelli R, Momah DU, Wahab S, Kim RS, Norman M, Zhang E, Hasoon J, Orhurh V, Viswanath O, Yazdi C, Chen GH, Simopoulos TT, Gill J. Pain Scales: What Are They and What Do They Mean. Curr Pain Headache Rep. 2024 Jan;28(1):11-25. doi: 10.1007/s11916-023-01195-2. Epub 2023 Dec 7. PMID 38060102
- [Background] Wells G, Becker JC, Teng J, Dougados M, Schiff M, Smolen J, Aletaha D, van Riel PL. Validation of the 28-joint Disease Activity Score (DAS28) and European League Against Rheumatism response criteria based on C-reactive protein against disease progression in patients with rheumatoid arthritis, and comparison with the DAS28 based on erythrocyte sedimentation rate. Ann Rheum Dis. 2009 Jun;68(6):954-60. doi: 10.1136/ard.2007.084459. Epub 2008 May 19. PMID 18490431
- [Background] Kim J, Kim I, Kim YE, Koh SB. The Four Square Step Test for Assessing Cognitively Demanding Dynamic Balance in Parkinson's Disease Patients. J Mov Disord. 2021 Sep;14(3):208-213. doi: 10.14802/jmd.20146. Epub 2021 May 26. PMID 34030434
- [Background] Kocaman H, Canli M, Alkan H, Yildirim H, Yildiz NT. The Reliability and Validity of the Modified Four Square Step Test in Individuals with Anterior Cruciate Ligament Reconstruction. Indian J Orthop. 2023 Sep 13;57(11):1819-1825. doi: 10.1007/s43465-023-00993-5. eCollection 2023 Nov. PMID 37881277
- [Background] Horata ET, Eken F, Yesil M, Ozcan O. Validity and reliability of the modified four square step test in total HIP arthroplasty. J Bodyw Mov Ther. 2024 Oct;40:345-349. doi: 10.1016/j.jbmt.2024.04.028. Epub 2024 Apr 16. PMID 39593608
- [Background] Verma A, Samuel AJ, Aranha VP. The four square step test in children with Down syndrome: Reliability and concurrent validity. J Pediatr Neurosci. 2014 Sep-Dec;9(3):221-6. doi: 10.4103/1817-1745.147573. PMID 25624923
- [Background] Aldirmaz E, Ugur F, Yilmaz O, Karaduman A, Alemdaroglu-Gurbuz I. A New Instrument to Assess Dynamic Balance in Children with Duchenne Muscular Dystrophy: Four Square Step Test and Its Validity, Reliability and Feasibility. Dev Neurorehabil. 2023 Jan;26(1):27-36. doi: 10.1080/17518423.2022.2143924. Epub 2022 Nov 11. PMID 36367327
- [Background] Tanrıöğer Soyuer F. Valıdıty And Relıabılıty Of "Four-Square Step Test" In Adolescent Cerebral Palsy2018.
- [Background] Taylor S, Pemberton S, Barker K. Validity of the four-square step test in persons with haemophilia. Haemophilia. 2022 Mar;28(2):334-342. doi: 10.1111/hae.14482. Epub 2022 Jan 12. PMID 35020243
- [Background] Toprak CS, Duruoz MT, Gunduz OH. Static and Dynamic Balance Disorders in Patients With Rheumatoid Arthritis and Relationships With Lower Extremity Function and Deformities: A Prospective Controlled Study. Arch Rheumatol. 2018 Jan 15;33(3):328-334. doi: 10.5606/ArchRheumatol.2018.6720. eCollection 2018 Sep. PMID 30632523
- [Background] Aydog E, Bal A, Aydog ST, Cakci A. Evaluation of dynamic postural balance using the Biodex Stability System in rheumatoid arthritis patients. Clin Rheumatol. 2006 Jul;25(4):462-7. doi: 10.1007/s10067-005-0074-4. Epub 2005 Oct 25. PMID 16247584
- [Background] Wasserman A. Rheumatoid Arthritis: Common Questions About Diagnosis and Management. Am Fam Physician. 2018 Apr 1;97(7):455-462. PMID 29671563
- [Background] Wu D, Li Y, Xu R. Can pyroptosis be a new target in rheumatoid arthritis treatment? Front Immunol. 2023 Jun 22;14:1155606. doi: 10.3389/fimmu.2023.1155606. eCollection 2023. PMID 37426634
- [Background] Yetis M, Kocaman H, Canli M, Alkan H, Yildirim H, Yildiz NT, Kuzu S. Validity and reliability of the Modified Four Square Step Test in individuals with ankle sprain. J Orthop Surg Res. 2024 Mar 15;19(1):182. doi: 10.1186/s13018-024-04664-5. PMID 38491530
- [Background] Smolen JS, Aletaha D, McInnes IB. Rheumatoid arthritis. Lancet. 2016 Oct 22;388(10055):2023-2038. doi: 10.1016/S0140-6736(16)30173-8. Epub 2016 May 3. PMID 27156434